CLINICAL TRIAL: NCT00693771
Title: A Prospective Study to Optimize Insulin Treatment by Basal Regimen With Insulin Glargine in Type-2-Diabetic Patients Previously Uncontrolled on Premixed Insulin
Brief Title: Study to Optimize Insulin Treatment by Basal Regimen With Insulin Glargine in Type-2-Diabetic Patients Previously Uncontrolled on Premixed Insulin
Acronym: OPTIMIZATION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_02756
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — Once daily and up-titrate accordingly

SUMMARY:
Primary objective:

To show an improvement in HbA1c control after 4 months of treatment with insulin glargine + Oral Anti Diabetic (OAD) in patients previously uncontrolled on premixed insulin (with OAD)

Secondary objective:

Improvement of Fasting blood glucose (FPG) after 4 months treatment (% of patients treated to target HbA1c ≤7.0% and/or FBG≤6.0mmol/L). Frequency of hypoglycemic episodes, quality of life with basal+ OAD regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus inadequately controlled at least 3 months on premixed insulin with 1 or 2 OADs
* 7.5 ≤ HbA1c ≤ 9.5%
* FPG ≥6.7 mmol/L
* History of Diabetes mellitus ≤10 years
* Premix insulin daily dosage ≤ 50 IU/Day

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Former treated on TZD
* Pregnancy / Lactation
* Creatine ≥1.5 mg/dl
* Hepatic disease, jaundice,or ALT/AST≥ 2.5 times of normal range
* Hormone therapy,
* Acute status of Diabetes complications
* Severe concomitant disease or complications with high risk of unexpected fatal events, like Myocardial Infarct, stroke, heart failure.
* Allergic to insulin glargine or any ingredient
* Participation in another clinical trial within 3 months

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
HbA1c values | At baseline and 16 weeks

SECONDARY OUTCOMES:
Adverse events including hypoglycemia | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rui Yan Ding, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China

REFERENCES:
- [Derived] Yang W, Du J, Zhang M, Hou J, Zhang X, Cui N. Predictors of HbA1c reduction and hypoglycemia in type 2 diabetes mellitus individuals switching from premixed to basal insulin: an exploratory analysis of optimization study. Curr Med Res Opin. 2022 Nov;38(11):1807-1814. doi: 10.1080/03007995.2022.2105538. Epub 2022 Aug 9. PMID 35943899